CLINICAL TRIAL: NCT06295094
Title: The Efficacy of Pressurised Intraperitoneal Aerosol Chemotherapy (PIPAC) Combined With CURativE Intent Minimally Invasive Radical Resection in High-risk Gastric Cancer Patients. A Multicentre, Randomised, Open-label Phase-II Study
Brief Title: The Efficacy of PIPAC and Minimally Invasive Radical Resection in High-risk Gastric Cancer Patients.
Acronym: EPICURE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIPAC-OPC6
Record Dates: First submitted 2024-02-19; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer; Chemotherapy, Adjuvant; Peritoneal Metastases; Minimally Invasive Surgical Procedures
Keywords: PIPAC; Gastric cancer; Minimally invasive gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pressurized intraperitoneal chemotherapy (PIPAC) (Experimental): In the intervention arm, conventional pressurized intraperitoneal chemotherapy (PIPAC) with cisplatin (10.5 mg/m2 body surface in 150ml saline) and doxorubicin (2.1 mg/m2 body surface in 50ml saline) is performed through Medical Device Regulation (MDR) class IIb the CE-certified nebuliser by certified PIPAC surgeons directly after the completion of the minimally invasive gastric resection and reconstruction using the remaining relevant ports. Chemotherapy is administered through a CE-certified nebulizer according to the manufacturer's manual and followed by 30 minutes of simple diffusion. The carbondioxide is evacuated through a closed system, and the abdominal wall is closed according to local surgical standards.
  The same procedure is repeated, incorporating the same compounds and dose regimens six to eight weeks postoperatively and before the start of the adjuvant part of the perioperative systemic chemotherapy.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin
- Standard (No Intervention): In the control arm, patients will undergo minimally invasive D2 gastrectomy

INTERVENTIONS:
Drug: Cisplatin — 10.5 mg/m2 body surface in 150ml saline
  Arms: Pressurized intraperitoneal chemotherapy (PIPAC)
Drug: Doxorubicin — 2.1 mg/m2 body surface in 50ml saline
  Arms: Pressurized intraperitoneal chemotherapy (PIPAC)

SUMMARY:
The goal of this randomized clinical trial is to investigate whether pressurized intraperitoneal chemotherapy (PIPAC), delivered immediately after minimally invasive D2 gastrectomy and repeated 6-8 weeks later, improves 12-month peritoneal disease-free survival in patients with high-risk gastric adenocarcinoma when compared to standard treatment.

DETAILED DESCRIPTION:
Despite declining incidence, gastric adenocarcinoma (GAC) is considered the fifth most common cancer worldwide and the third leading cause of cancer death globally. Its incidence varies across different parts of the globe, with a low incidence in the West. In East Asia, especially Japan and Korea, the incidence of distal GAC remains high, whereas proximal GAC tends to dominate in the West. Gastroesophageal junction (GEJ) adenocarcinomas that have the epicentre in the proximal 2 to 5 cm of the stomach (Siewert type III) should be staged and treated as GAC.

The consensus in most Western countries is that medically fit GAC patients should undergo D2 gastrectomy, carried out in specialised, high-volume centres with perioperative outcomes in terms of morbidity and mortality rates comparable to those presented in Japan and South Korea. A minimally invasive D2 gastrectomy has emerged as a valid and preferable alternative to open surgery.

Despite significant progress in implementing preventive strategies and curative treatment of premalignant and early neoplastic gastric lesions, most GAC patients still present with advanced stages of the disease, leading to a dismal prognosis even after treatments with curative intent. Given that many patients relapse following surgery, various multimodal treatment strategies have been studied to improve survival rates, mainly by combining surgery with systemic treatment in the form of perioperative chemotherapy. Clinical research has explored and documented the concept of perioperative chemotherapy in GAC and cancers originating in the distal esophagus and GEJ. Noteworthy is that some of these have suggested that the tumours with the most obvious responses to corresponding regimens originate in the esophagus and GEJ. Moreover, GACs of poorly differentiated tubular type or poorly cohesive cancer, regardless the presence of signet-ring cells type has been reported to be more resistant to chemotherapy regimens. Another observation with clinical implications is that GAC patients with malignant cells retrieved from peritoneal lavage before surgery have an extremely poor prognosis. Hence, laparoscopy with peritoneal lavage for malignant cells is recommended in all stage IB-III gastric cancers, otherwise considered potentially resectable, to exclude radiologically occult metastatic disease. The true value of this information may be even greater for patients with T3/T4 disease. Considering the above-mentioned challenges, it is critically important to explore novel multimodal therapeutic concepts in GAC since current therapeutic strategies offer these patients a limited option for cure.

The occurrence of peritoneal metastases (PM) has a significant negative impact on the overall prognosis, with a median survival of three to four months without treatment. None of the available chemotherapy regimens has reduced or prevented the risk of PM. It is commonly believed that PM occur through the deposition of tumour cells either by the direct extension and subsequent cellular exfoliation or through the traumatic dissemination of cancer cells during surgery. Clinical validation of the concept of direct spread is also provided by observing the higher rate of PM seen with increasing tumour stages (T-stages) and serosal involvement. This is also supported by the association of between positive peritoneal cytology and a higher tumour stage.

Sixty percent of lavage cytology-negative patients will convert to a cytology-positive state immediately after gastrectomy. Accordingly, it can be argued that during gastrectomy, cancer cells within the dissected lymphatic channels and blood vessels are released to and disseminated throughout the abdominal cavity. Free cancer cells can then attach to the peritoneal surface, a process facilitated by the action of cytokines and the deposition of fibrin layers, allowing for the entrapment of those cells. This new restrictive-peritoneal environment is thought to hinder the penetrance of cytotoxic drugs delivered systemically and provides grounds for the launch of intraperitoneal treatments.

Based on the minimal effects of traditional regimens on GAC, exploring alternative perioperative therapeutic concepts appears of the highest clinical significance. Since only a fraction of the systemically administered chemotherapy reaches the peritoneum, the effect of intraperitoneal chemotherapy has been extensively studied. A new aerosol technique, Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC), improves intraperitoneal delivery and subsequent uptake of chemotherapy. It has shown promising results in patients with PM from colorectal, ovarian, pancreatic, and gastric cancer. Furthermore, PIPAC is feasible, safe, and well tolerated by many patients when administered in the palliative setting.

Randomised studies on prophylactic treatment of high-risk GAC patients (serosal invasion) using intraperitoneal chemotherapy or hyperthermic intraperitoneal chemotherapy (HIPEC) are mainly from Asian institutions. The risk of postoperative morbidity and mortality did not seem to be negatively influenced by intraoperative, intraperitoneal chemotherapy, contrasting to western non-randomized trials reporting considerable morbidity and mortality after these combined procedures. Thus, the use of prophylactic HIPEC in non-metastatic high-risk GAC is still debated.

Data from Odense PIPAC Centre on the outcome of PIPAC with low-dose cisplatin and doxorubicin in GAC patients with chemotherapy-resistant PM revealed objective tumour response in 40% of the patients after three PIPAC directed therapies. An additional 20% had no further tumour progression. These observations in GAC patients deliver further evidence suggesting that PIPAC can induce regression of resistant PMs in several cancer types and carries the potential to meet the clinical need for new and better therapies. Our results also provide evidence that low-dose PIPAC therapy might effectively treat patients with recurrent, chemo-resistant gastric PMs, including the poorly differentiated tubular type or poorly cohesive cancer.

The pivotal question is whether PIPAC delivered immediately after a laparoscopic D2 gastrectomy for GAC can reduce the risk of recurrent PM. Our institutions' recent phase I trial has shown this therapeutic concept to be feasible and safe. Hence, a randomised phase-II clinical trial must be conducted to assess the impact of PIPAC on disease-free survival in patients with high-risk GAC who are offered surgical treatment with curative intent.

ELIGIBILITY:
Inclusion criteria

* Gastric or Gastroesophageal junction Siewert type III adenocarcinomas
* Clinical T3-4a-stages

  1. Any differentiation grade
  2. Any histological subtype
* Clinical T2-stage

  a. If poorly differentiated or of the poorly cohesive histological subtype, with or without the presence of signet-ring cells
* Any clinical T-stage with positivity for malignant cells on abdominal lavage cytology, which is converted to cytology negative in response to neoadjuvant chemotherapy.
* Any clinical nodal-stage
* clinical M0-stage (positive abdominal wash cytology, which is converted to cytology negative in response to neoadjuvant therapy, is permitted)
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-1
* Age 18 - 80 years
* Undergoing robotic or laparoscopic D2 gastrectomy
* Able and willing to provide written informed consent and to comply with the clinical study protocol
* Fertile women must have a negative pregnancy test at the time of inclusion and must use adequate contraception.

Exclusion criteria

* Previous allergic reaction to cisplatin, doxorubicin or other platinum-containing compounds.
* Renal impairment, defined as glomerular filtration rate (GFR) < 40 ml/min (Cockcroft-Gault Equation).
* Myocardial insufficiency, defined as New York Heart Association (NYHA) class 3-4.
* An impaired liver function, defined as bilirubin ≥ 1.5 x upper normal limit (UNL).
* An inadequate haematological function, defined as absolute neutrophil count (ANC) <1.5 x 109/l and platelets <100 x 109/l.
* Any other condition or therapy which, in the investigator's opinion, may pose a risk to the patient or interfere with the study objectives.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Peritoneal disease-free survival | 12 months
  Peritoneal disease-free survival (P-DFS) defined as no signs of peritoneal recurrence on (PET) CT and/or control laparoscopy with at least 12 months follow-up after minimally invasive D2-gastrectomy

SECONDARY OUTCOMES:
Disease-free survival | 12 months
  Rate of disease-free survival (DFS) with at least 12 months of follow-up
Overall survival | 12 months
  Rate of overall survival with at least 12 months of follow-up
Length of stay | 30 days
  Length of stay (LOS) (Surgery = Day 0)
Postoperative toxicity | 30 days
  Rate of patients with 30 days postoperative toxicity (CTCAE)
Postoperative complications | 30 days
  Rate of patients with 30 days postoperative complications (Dindo-Clavien)
Postoperative mortality | 90 days
  Rate of patients with 90 days postoperative mortality
Rate of positive peritoneal lavage | 90 days
  Rate of positive peritoneal lavage at surgery
Patient-reported Quality of life | 30 days & 12 months
  European Organisation for Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Patient-reported Quality of life | 30 days & 12 months
  European Organisation for Treatment of Cancer Quality of Life Questionnaire Gastric Cancer (EORTC QLC-STO22)
Number of patients not receiving adjuvant chemotherapy | 90 days
  Number of patients not receiving adjuvant chemotherapy as planned due to PIPAC related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bau Mortensen, DMSci, PhD, Study Director — University of Southern Denmark (sdu.dk)
Locations (5):
- City of Hope, Duarte, California, United States
- Odense University Hospital, Odense C, Denmark
- University Hospital Lille, Lille, France
- Charité, University of Berlin, Berlin, Germany
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No